CLINICAL TRIAL: NCT05471856
Title: Phase Ia, First in Human Open Label Dose Escalation Trial Evaluating Intravenous BI 1703880 in Combination With Intravenous Ezabenlimab for Treatment of Advanced Solid Tumours
Brief Title: A Study to Test How Different Doses of BI 1703880 in Combination With Ezabenlimab Are Tolerated in People With Different Types of Advanced Cancer (Solid Tumours)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1480-0001; 2022-000298-22 (EudraCT Number); U1111-1303-5359 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP)); 2024-511501-37-00 (EU CTIS Number)
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BI 1703880 (Cycle 1) then BI 1703880 + ezabenlimab (Cycle 2 onwards) (Experimental)
  Interventions: Drug: BI 1703880; Drug: Ezabenlimab

INTERVENTIONS:
Drug: BI 1703880 — BI 1703880
Drug: Ezabenlimab — Ezabenlimab
  Other Names: BI 754091

SUMMARY:
This study is open to adults with different types of advanced cancer. People can take part if previous treatment was not successful, or no treatment exists.

The purpose of this study is to find the highest dose of a medicine called BI 1703880 that people with advanced cancer can tolerate when taken together with ezabenlimab.

BI 1703880 and ezabenlimab are medicines that may help the immune system fight cancer. In this study, BI 1703880 is given to people for the first time.

Participants get BI 1703880 and ezabenlimab as infusions into a vein. During the first 6 weeks, they get BI 1703880 once a week. Later, they get BI 1703880 every 3 weeks. After the first 3 weeks, they get ezabenlimab in addition every 3 weeks.

Participants can get BI 1703880 for up to 1 year and ezabenlimab for up to 2 years as long as they benefit from treatment and can tolerate it. During this time, they visit the study site regularly. At these visits, the doctors check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of an advanced, unresectable and/or metastatic or relapsed/refractory solid tumour. Patient must have at least one measurable lesion (according to Response Criteria in Solid Tumours (RECIST 1.1)).
* Patient must have exhausted or refused established treatment options for the malignant disease, or is not eligible for established treatment options.
* Has a lesion amenable to pre-treatment and on-treatment biopsy and patient consents to both biopsies.
* Medically fit and willing to undergo all mandatory trial procedures.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
* Adequate organ function or bone marrow reserve as demonstrated at screening by the following laboratory values:

  * Absolute neutrophil count ≥ 1.5x10^9/L (≥ 1.5x10^3/μL, ≥ 1500/mm3); platelet count ≥ 100x10^9/L (≥ 100x10^3/μL, ≥ 100x10^3/mm3), without the use of hematopoietic growth factors within 4 weeks of start of trial medication
  * Haemoglobin ≥ 90 g/L (≥ 9.0 g/dL, ≥ 5.6 mmol/L)
  * Estimated glomerular filtration rate (eGFR) ≥60 ml/min/1.73m^2 (as determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula)
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 x ULN if no demonstrable liver metastases, or otherwise ≤ 5 x ULN if transaminase elevation is attributable to liver metastases.
  * Total bilirubin ≤ 1.5 x ULN, except for patients with Gilbert's syndrome: total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
  * partial thromboplastin time (PTT) / activated partial thromboplastin time (aPTT) <1.5 x ULN
* Patients ≥18 years of age or over the legal age of consent in countries where that is greater than 18 years at the time of signature of the informed consent form (ICF).
* Signed and dated written ICF in accordance with International Council for Harmonisation- Good Clinical Practice (ICH-GCP) and local legislation, obtained before performing any protocol related procedures that are not part of normal standard of practice care. Note: If a patient declines to participate in the voluntary biobanking component of the trial, he/she will not be excluded from other aspects of the trial.

Further inclusion criteria apply

Exclusion Criteria:

* Any investigational or antitumour treatment within 4 weeks or 5 half-life periods prior to the first treatment whichever is shorter.
* Prior STING agonist therapy.
* Prior intolerability of a anti-programmed cell death protein 1 (PD-1) or anti-programmed cell death ligand 1 (PD-L1) therapy.
* History of allergy or hypersensitivity to study agent components.
* Immunosuppressive therapies including, but not limited to, systemic corticosteroids at doses exceeding >10 mg/day of prednisone or equivalent, and tumour necrosis factor-alpha blockers.
* Persistent toxicity from previous treatments (including immune related Adverse Events (irAEs)) that has not resolved to Grade ≤1, except for alopecia, xerostomia, and immunotherapy related endocrinopathies.
* Evidence of active, non-treatment related autoimmune disease, except for endocrinopathies.
* History or complication of pneumonitis or interstitial lung disease within the last 12 months, or any prior pneumonitis related to immunotherapy.

Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2028-09-13 (Estimated); Study Completion 2028-09-13 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities (DLTs) during the maximum tolerated dose (MTD) evaluation period | up to 6 weeks

SECONDARY OUTCOMES:
Occurrence of DLTs during the on-treatment period | up to 804 days
Maximum measured concentration of BI 1703880 in plasma (Cmax) | up to 804 days
Area under the concentration-time curve of BI 1703880 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 804 days

CONTACTS AND LOCATIONS:
Locations (13):
- United States (3):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - John Theurer Cancer Center, Hackensack, New Jersey
- Japan (3):
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Saitama Medical University International Medical Center, Saitama, Hidaka
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- Spain (4):
  - Hospital Universitari Vall D Hebron, Barcelona
  - CIO Clara Campal, Madrid
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clinico Universitario De Valencia, Valencia
- United Kingdom (3):
  - The Royal Marsden Hospital, Chelsea, London
  - Churchill Hospital, Oxford
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Harrington K, Kitano S, Gambardella V, Parkes EE, Moreno I, Alonso G, Doi T, Berz D, Gutierrez ME, Fernandez N, Schmohl M, Barrueco J, LoRusso P. Open-label, phase Ia study of STING agonist BI 1703880 plus ezabenlimab for patients with advanced solid tumors. Future Oncol. 2025 Jan;21(2):195-200. doi: 10.1080/14796694.2024.2441107. Epub 2025 Jan 16. PMID 39817655
- See also: Related Info — http://www.mystudywindow.com